CLINICAL TRIAL: NCT01949207
Title: Randomised Controlled Study to Determine Whether Treating Incompetent Perforating Veins at the Time of Endothermal Varicose Vein Surgery for Truncal Reflux Reduces Recurrence After Varicose Vein Treatments.
Brief Title: RCT - Does Treating Incompetent Perforators Reduce Recurrence?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT20133
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Varicose Veins
Keywords: Incompetent perforating veins; EVLA; Phlebectomies; TRansluminal Occlusion of Perforators (TRLOP) closure of incompetent perforators.
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVLA, phlebectomies & Trlop closure of incompetent perforators (Experimental): endovenous laser ablation (EVLA) of great saphenous vein (GSV) plus phlebectomies plus TRansluminal Occlusion of Perforators (TRLOP) closure of incompetent perforators.
  Interventions: Procedure: EVLA; Procedure: phlebectomies; Procedure: TRansluminal Occlusion of Perforators (TRLOP)
- EVLA & phlebectomies (Experimental): endovenous laser ablation (EVLA) of great saphenous vein (GSV) + phlebectomies.
  Interventions: Procedure: EVLA; Procedure: phlebectomies

INTERVENTIONS:
Procedure: EVLA — Endovenous laser ablation of great saphenous vein
Procedure: phlebectomies — removal of incompetent veins
Procedure: TRansluminal Occlusion of Perforators (TRLOP) — TRansluminal Occlusion of Perforators (TRLOP) closure of incompetent perforators.
  Arms: EVLA, phlebectomies & Trlop closure of incompetent perforators

SUMMARY:
The aim of this randomised case-controlled trial is to investigate whether ablation of incompetent perforating vein in addition to ablation of truncal vein reduces the rate of recurrent varicose veins post-treatment compared with patients who only have ablation of the truncal vein, who are left with untreated incompetent perforating veins.

ELIGIBILITY:
Inclusion Criteria:

* Primary varicose veins caused by great saphenous vein reflux
* At least one incompetent perforating vein refluxing into the varicosities
* Over 18 years of age

Exclusion Criteria:

* Reflux from pelvic vein origin or small saphenous vein
* Previous varicose vein surgery,
* Incompetent perforators remote from the varicosities treated,
* Deep vein incompetence
* Deep vein obstruction or occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Differences in the level of significant recurrence between the two treatment pathways | Four weeks, three months, six months, one year, two years, three years, four years and five years post-surgery
  Differences in the level of significant recurrence between the two treatment pathways at each follow up.
  Significant recurrence would be indicated if the participant demonstrates varicose veins greater than 3mm in diameter, varicose veins associated with thrombophlebitis or skin changes such as venous eczema, red skin or brown skin overlying the veins which require further treatment.

SECONDARY OUTCOMES:
Differences in insignificant recurrence between the two treatment pathways | Four weeks, three months, six months, one year, two years, three years, four years and five years post-surgery
  Evidence of insignificant recurrence - thread veins, reticular veins or varicose veins less than 3mm in diameter.
Patient reported symptom severity | Four weeks, three months, six months, one year, two years, three years, four years and five years post-surgery
  Patient reported symptom severity - the Aberdeen questionnaire
Patient reported quality of life | Four weeks, three months, six months, one year, two years, three years, four years and five years post-surgery
  Patient reported quality of life - The Chronic Venous Insufficiency Questionnaire (CIVIQ)
Patient satisfaction with treatment. | Four weeks, three months, six months, one year, two years, three years, four years and five years post-surgery
Clinician reported severity of symptoms | Four weeks, three months, six months, one year, two years, three years, four years and five years post-surgery
  CEAP and VCCS scores

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, Professor, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom